CLINICAL TRIAL: NCT06705270
Title: Randomized Controlled Trial Comparing the Impact of Patient Education Strategies on the Antidepressant Response to Propofol Sedation
Brief Title: Sedation and Guided Education for Depression Study
Acronym: SAGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Theresa Lii, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 76737
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2025-05-19 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Propofol; Sedation; Patient education; Antidepressant; Major depressive disorder; Electroencephalography
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Response-focused education (Active Comparator): Patient education that is focused on treatment response
  Interventions: Behavioral: Response-focused education
- Diagnosis-focused education (Active Comparator): Patient education that is focused on the diagnosis of major depressive disorder
  Interventions: Behavioral: Diagnosis-focused education

INTERVENTIONS:
Behavioral: Response-focused education — Once participants recover from sedation, they will receive education that is focused on their response to treatment.
  Arms: Response-focused education
Behavioral: Diagnosis-focused education — Once participants recover from sedation, they will be provided education that is focused on their diagnosis of major depressive disorder.
  Arms: Diagnosis-focused education

SUMMARY:
The goal of this clinical trial is to understand how patient education surrounding a one-time, consciousness-altering medical intervention impacts the antidepressant response to the intervention in adults with major depressive disorder. In this study, the consciousness-altering medical intervention is a single infusion of propofol, an intravenous anesthetic which might have antidepressant properties.

The main question this study aims to answer is: Does the focus of patient education influence the antidepressant response to a single intravenous infusion of propofol?

Researchers will compare response-focused vs. diagnosis-focused education.

Qualifying participants will:

* Undergo a single intravenous infusion of propofol which will induce a temporary state of sedation
* Wear an EEG cap that records brain activity during sedation
* Be randomized to receive either response-focused or diagnosis-focused education about their brain signals after they recover from sedation
* Be asked to fill out surveys about their mood and other measures of well-being before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder of at least moderate severity
* Able to read, understand, and provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Certain substance use disorders
* Daily use of opioids and/or benzodiazepines
* History of psychosis, schizophrenia, or schizoaffective disorder
* Body mass index greater than 35 kg/m2
* Obstructive sleep apnea that is moderate and untreated, or severe
* Any gastrointestinal condition placing the patient at significant risk of aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Depression severity | From enrollment to 28 days after treatment
  The 16-item Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR-16) assesses the severity of depressive symptoms experienced by an individual. Items are self-rated on a 4-point scale tailored to each depression symptom. Higher total scores indicate greater depression severity.

OTHER OUTCOMES:
Sedation awareness | Immediately upon recovery from sedation
  The modified Brice Questionnaire will be used to evaluate what the participant remembers between the time of induction and their awakening from sedation.
Participant expectations | From enrollment to 28 days after treatment
  Participants will be asked to rate how effective they expect their treatment to be on a scale from 0 (not effective at all) to 100 (completely effective) and indicate the amount of confidence they have on a scale from 0% to 100%.
Sleep disturbance | From enrollment to 28 days after treatment
  The 8-item PROMIS Sleep Disturbance Short Form assesses an individual's perception of their sleep quality. Items are self-rated on a 5-point scale ranging from 1 ("Not at all") to 5 ("Very much"). Raw scores are converted to standardized T-scores, with higher a T-score representing more severe sleep disturbance.
Anxiety symptoms | From enrollment to 28 days after treatment
  The 7-item Generalized Anxiety Disorder (GAD-7) Scale assesses the severity of anxiety symptomsover the past two weeks. Items are self-rated on a 4-point scale ranging from 0 ("Not at all") to 3 ("Nearly every day"), reflecting the frequency of symptoms. Higher total scores indicate greater anxiety symptom severity.
Anhedonia | From enrollment to 28 days after treatment
  The 14-item Snaith-Hamilton Pleasure Scale (SHAPS) measures an individual's capacity to experience pleasure from various activities over the past two weeks, the absence of which indicates anhedonia. Items are self-rated on a 4-point scale ranging from 0 ("Strongly disagree") to 3 ("Strongly agree"). Lower total scores indicate greater degree of anhedonia.
Peace of mind | From enrollment to 28 days after treatment
  The 7-item Peace of Mind Scale assesses an individual's overall sense of inner calm and contentment. Items are self-rated on a 5-point scale ranging from 1 ("Not at all") to 5 ("All of the time"). Higher total scores reflect a greater sense of peace of mind.
Emotion regulation | From enrollment to 28 days after treatment
  The 10-item Emotion Regulation Questionnaire (ERQ) assesses individual differences in the habitual use of cognitive reappraisal and expressive suppression strategies. Items are self-rated on a 7-point Likert scale. Higher scores on the cognitive reappraisal subscale indicate a greater tendency to reinterpret situations to manage emotions, while higher scores on the expressive suppression subscale indicate a greater tendency to inhibit outward emotional expression.
Frontal EEG theta power | Immediately before sedation start to time of recovery from sedation
  Electroencephalography (EEG) is a non-invasive technique that records electrical activity of the brain using electrodes placed on the scalp. Theta band (4 to 8 Hz) power in the frontal leads will be compared.
Adverse events | From treatment day to 28 days after treatment
  Safety will be assessed by tracking the number and severity of adverse events spontaneously reported by the participant and through surveillance of medical records (if available) by the research team. Suicidality will be specifically monitored using the Columbia Suicide Severity Rating Scale.

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, study outcomes, and data dictionaries
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Available upon request after publication of the trial's primary findings for up to 5 years.
Access Criteria: Researchers must submit a brief proposal and statistical analysis plan for review and approval by the investigators and execute a data sharing agreement.